CLINICAL TRIAL: NCT01963702
Title: Phase II Trial of Exploring the Predictive Factors of Docetaxol Plus Capecitabine(TX) Regimen and Oxaliplatin Plus Capecitabine (XELOX) Regimen in the First Line Treatment of Patients With Metastatic Gastric Cancer (MGC)
Brief Title: A Phase II Trial of Exploring the Predictive Factors of TX and XELOX Regimen in the First Line Treatment of MGC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaodong Zhu, associate professor, Fudan University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FDZL-TXELOX
Record Dates: First submitted 2013-10-09; First posted 2013-10-16 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Gastric Cancer
Keywords: predictive factor; response; gastric neoplasm; oxaliplatin; docetaxol; capecitabine
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Docetaxol ＆Capecitabine (TX) (Experimental): Docetaxol: 75 mg/m2 d1, (From MAY 15th 2013, the dose was reduced to 60mg/m2 for high incidence of G3/4 myelosuppression after approved by institute Ethics Committee) ; Capecitabine 1000 mg/m2 bid ×14d; Repeat every 3 weeks, until disease progression or intolerable toxicity or patients withdrawal of consent,or total 8 cycles
  Interventions: Drug: Docetaxol; Drug: Capecitabine
- Oxaliplatin ＆Capecitabine (XELOX) (Active Comparator): Oxaliplatin: 130 mg/m2 d1; Capecitabine 1000 mg/m2 bid ×14d; Repeat every 3 weeks, until disease progression or intolerable toxicity or patients withdrawal of consent,or total 8 cycles
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Docetaxol
  Arms: Docetaxol ＆Capecitabine (TX)
Drug: Oxaliplatin
  Arms: Oxaliplatin ＆Capecitabine (XELOX)
Drug: Capecitabine
  Other Names: xeloda

SUMMARY:
Platinum, fluorouracil and taxane based regimen are all acceptable in the first line treatment of metastatic gastric cancer. The TX and XELOX regimen are two common regimen used in MGC. whichever regimen is used, the average response rate is less than 50%. So a rather part of patients can't get benefit from the treatment. It is urgent to find out the predictive factors of these regimens in order to get a higher response and better survival outcome.

DETAILED DESCRIPTION:
Patients with MGC will be treated with TX or XELOX regimen. Before treatment, 14 days after treatment and after progression, the blood sample will be collected. Primary tumor blocks will also of collected. These samples will be used to detect predictive factors of the two types first line therapy.

ELIGIBILITY:
Inclusion Criteria:

* Chemo-naive patients with metastatic, unresectable, histologically confirmed gastric or Gastroesophageal adenocarcinoma; Patients who received adjuvant chemotherapy, the duration from the last therapy to relapse at least longer than 6 months
* Patient must have at least one measurable lesions (RECIST 1.1)
* 18 Years to 75 years
* Written informed consent obtained
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Patients must have adequate organ and marrow function as defined below:
* neutrophilicgranulocyte greater than/equal to 1,500/mm3;
* platelets greater than/equal to 90,000/ mm3;
* hemoglobin greater than/equal to 9 gm/dL (may be transfused to maintain or exceed this level);
* total bilirubin less than/equal to 1.5 within institutional upper limit of normal (IULN);
* Aspartate Transaminase (AST,SGOT)/Alanine transaminase (ALT,SGPT) less than/equal to 2.5 times IULN
* serum creatinine less than/equal to 1.5 x IULN.

Exclusion Criteria:

* Active clinically serious infections (> grade 2 NCI-CTC version 3.0, National Cancer Institute-Common Terminology Criteria for Adverse Events)
* Symptomatic metastatic brain or meningeal tumors
* History of organ allograft
* Patients undergoing renal dialysis
* chronic inflammatory bowel disease; ileus; genetic fructose intolerance
* Patients who received adjuvant chemotherapy and the duration from the last therapy less than 6 months
* Receive previously radiotherapy in measurable regions
* Pregnancy or lactating status
* Concurrent malignancy other than nonmelanoma skin cancer, or in situ cervix carcinoma
* Clinically relevant coronary artery disease or history of a myocardial infarction within the last 12 months
* Acute or subacute intestinal occlusion or history of the inflammatory bowel disease
* Any factors that influence the usage of oral administration

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
objective response | 6 weeks
  RECIST 1.1 (Response Evaluation Criteria in Solid Tumors) will be used to evaluate the response of each patient every 6 weeks. The main purpose of this study is to search for the biomarkers which will predict the response of patients with MGC received TX or XELOX regimen as first line therapy

SECONDARY OUTCOMES:
progression free survival (PFS) | From randomization until first documented progression or date of death from any cause, whichever came first (up to 60 months)
  PFS is defined as from the date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months

OTHER OUTCOMES:
overall survival(OS) | from the date of randomization until the date of death from any cause, assessed up to 60 months
  OS is defined as from the date of randomization until the date of death from any cause, assessed up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, M.D / Ph.D, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China